CLINICAL TRIAL: NCT05566925
Title: Patients' Perceptions of Assessment and Treatment of Knee Osteoarthritis on the First Visit in Primary Care - a Qualitative Study
Brief Title: Patients' Perceptions of Assessment and Treatment of Knee Osteoarthritis in Primary Care
Status: Active, not recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 276518_interview_KOA
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Perception; Experience; Physiotherapist; Triage; Direct access
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Restraint, Physical; Therapeutics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Direct access to physiotherapist for assessment, diagnosis and treatment. — Patients with knee osteoarthritis will be interviewed about their experience of being assessed, diagnosed and treated by a physiotherapist first in primary care.

SUMMARY:
Background: To diagnose osteoarthritis (OA), Swedish guidelines recommend an overall assessment including patient history, symptoms, and clinical findings. However, diagnostic radiography is not recommended when assessing OA. Assessing and giving core treatments of patients with knee OA (KOA) is included in physiotherapists' area of expertise. Former studies show that there is no statistically significant difference in health-related quality of life for patients with KOA assessed by physiotherapists compared to being assessed by a physician in primary care. There is also research showing that costs can be reduced with a physiotherapist as first assessor. A task-shifting care model with physiotherapists as the primary assessor, can result in a reduced waiting time to recommended treatment for patients with KOA, as well as increase the accessibility to physicians in primary care for patients with more severe health conditions.

Previous studies have explored expectations in patients with KOA and how they have experienced the health care when the first assessment and treatment has been performed by a physician. It has been described how referred patients with KOA have experienced physiotherapy treatment, and the physiotherapists' impact on exercise adherence. To the best of our knowledge, there are no studies describing how patients with KOA have experienced health care, when being referred directly to a physiotherapist for assessment and treatment.

The main purpose is to explore expectations, perceptions, and experiences among patients with KOA in primary care who have been assessed and treated by a physiotherapist. The second purpose is to explore the possible meaning of the first meeting when it comes to future self-care and experienced health status.

Methods: Estimated 12-15 patients with KOA will be recruited from rehabilitation centers in Region Västra Götaland, Sweden, from October 2022 to February 2023. Semi-structured interviews will be conducted and will be analyzed with qualitative content analysis.

Expected results: This study is expected to contribute to a deeper understanding of what expectations patients with KOA have before they seek health care, how they experience physiotherapists as primary assessor in KOA and possible influences of the physiotherapy assessment and treatment on patients' perceived health after the rehabilitation period. This knowledge could be valuable when implementing new care models for patients with KOA.

DETAILED DESCRIPTION:
Background:

To diagnose osteoarthritis (OA), Swedish guidelines recommend an overall assessment with patient history, symptoms, and clinical findings, and diagnostic radiography is not recommended when assessing OA. The recommended core treatment should consist patient education, exercising, self-care and if necessary, weight loss, whereas assessing and giving core treatments of knee OA (KOA) is included in physiotherapists area of expertise. Former study show that there is no statistic significant difference in health-related quality of life for patients with KOA assessed by physiotherapists compared to being assessed by a physician in primary care. Furthermore, costs can be reduced with the model "physiotherapists first". A task-shifting care model with physiotherapists as the primary assessor can result in a faster track to recommended treatment for patients with KOA and increase the accessibility to physicians in primary care for patients with more severe health conditions.

Qualitative studies show that patients generally are skeptical to physiotherapists competence compared to physicians regarding assessing musculoskeletal disorders, and a physician assessment could be experienced as an assurance before being assessed and treated by physiotherapist. At the same time, one of these studies shows that there is an acceptance that advanced physiotherapy practitioner can be primary assessor for patients with musculoskeletal disorders. Previous patient experiences of physician assessment could affect patient's expectation of a physician to assess and diagnose their musculoskeletal disorder again, and a belief in need of further examinations with radiography could be another cause to consult a physician first.

Overall, patients with OA have had a negative view on conservative OA treatment and experienced that health care have trivialized their symptoms. Patients with KOA could feel hesitant to seek help due to beliefs of physicians' attitude regarding joint pain as a normal ageing symptom. This patient group have reported that their complaints were not taken seriously, and want more focus on the individual rather than the joint. Many patients assessed and treated by physicians report lack of understanding of OA and experience pain avoidance. Patients want other treatment options than drugs, and urge for more time for counselling and information about OA. Physicians experience difficulties in OA management due to time constraints, priorities, and in presenting and choosing treatments. Exercise was reported as an important factor in the management of OA. Referred patients with KOA treated with physiotherapy reported receiving treatments that was recommended for this patient group and the relationship between physiotherapists and patients are important for exercise adherence.

To the best of our knowledge, there are no studies of how patients with KOA, have experienced the health care, when being referred directly to a physiotherapist for assessment and treatment. To offer person-centred care for patients with suspected KOA, it is of value to get a deeper understanding of what expectations patients have and what possible meaning a primary assessment by physiotherapists have on patient's future self-care and experienced health status.

Purpose:

Firstly, the purpose is to explore expectations, perceptions, and experiences among patients with KOA who have sought primary care and being assessed and treated by a physiotherapist first. The second purpose is to explore the possible meaning of the first meeting when it comes to future self-care and experienced health status.

Question areas:

1. What expectations did patients with KOA have when they sought primary care for their knee pain? What was important before the first meeting with the health care?
2. How did patients with KOA experience their meetings with the health care?
3. Did the first meeting with health care influence the continued experience of health status for patients with KOA? If so, how?

Study design

Qualitative research study with an inductive approach. The consolidated criteria for reporting qualitative research' (COREQ) checklist will be used in the planning and reporting results of the study.

Patient recruitment and sample size

An estimation of 12-15 patients with diagnosed KOA will be recruited from rehabilitations centers in Region Västra Götaland, in southwestern Sweden, from October 2022 to February 2023. Patients will be recruited either by the physiotherapist who treated them, or through a search in a medical record database where patients with KOA will be contacted if they have been patients the last year on the rehabilitation centers. All participants will approve their participation through informed consent. The Swedish Ethical Review Authority have approved the study, reference number 2022-03479-01.

Data collection

Semi-structured interviews will be conducted by project leader CMHH. An interview guide will be designed and approved by the research group to ensure it answering to the purpose of the study. The interview guide will be pilot tested and approximately 1-2 interviews will be conducted. These interviews might be included in the analysis. The interviews are expected to last about 45-60 minutes and will be recorded with MP3-player or via the secure video conference call system. The interviewer will make a strategic selection of informants, to get a rich variation of the interview data. Data collection will end when no new information that corresponds to the purpose is added.

Participants will be strategically selected based on patient characteristics: gender, age, origin (born in Sweden or not), living alone or together with someone, educational level, pain duration, pain intensity, comorbidities, health care process. These data will be collected via questionnaires.

Data management

All data will be coded and managed according to the General Data Protection Regulation. All data will be confidential and only authorized will have access to the patient registry. No individual information can be identified since the results will be presented at group level. Data will be saved for at least 10 years to enable audit.

Analysis plan

Patient characteristics will be de-identified and presented on an individual level. The interview data will be listened through, and transcribed verbatim. A qualitative content analysis with inductive approach will be performed according to Graneheim and Lundman:

Initial phase: All interviews will be read thoroughly several times to get an overall feeling for the data. Data will be prepared in Microsoft Excel, Office 365 and thereafter transferred to the analytic data program NVivo Pro for Windows.

Analyzing the manifest content

First phase: Extracting meaning units based on the purpose. i.e., choosing contents that correspond to the purpose of the study.

Second phase: Condensing meaning units by shortening the texts without losing its context.

Third phase: Coding condensed meaning units. Labeling the content without losing the understanding or the relation to the context.

Analyzing the latent content

Fourth phase: Creating sub-/categories where codes with similar content will be sorted in as homogeneous internal and heterogeneous external categories as possible.

Fifth phase: If possible, the categories will be abstracted further to themes.

The project leader/first author (CMHH) will be responsible for transcribing, preparing and coding themes for all interviews. Preliminary categorizing and suggesting themes will also be conducted by CMHH. Every co-author (LN, LZ and CT) will read interviews and all authors will approve the analysis and its results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosed knee osteoarthritis, who have been assessed, diagnosed, and treated by a physiotherapist as primary assessor in primary care.
* The patient need to have had at least one month of treatment. The treatment period does not have to be finished.
* Assessed the last year
* Be able to understand and speak the Swedish language

Exclusion Criteria:

* Pregnancy
* Other severe psychic or somatic disorders or functional impairments that could have affected the treatment of knee osteoarthritis.
* Patient have had the interviewer as assessing and/or treating physiotherapist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with knee osteoarthritis in primary care who have been assessed, diagnosed and treated by a physiotherapist first.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Expectations before meeting with health care | From 1 to 12 months
  What expectations did patients with KOA have before meeting with health care? One of the question areas to be answered during a semi-structured interview.
Perceptions when meeting with health care | From 1 to 12 months
  What perceptions did patients with KOA have when meeting with the health care? One of the question areas to be answered during a semi-structured interview.
The meaning of the meetings with health care | From 1 to 12 months
  What possible influences did meetings with health care have on future self-care and health status? One of the question areas to be answered during a semi-structured interview.

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Mei Ho-Henriksson, PhD-student, Principal Investigator — Närhälsan, Region Västra Götaland
Locations (2):
- Sweden (2):
  - Närhälsan Lidköping Rehabmottagning, Lidköping, Västra Götaland County
  - Närhälsan Skara Rehabmottagning, Skara, Västra Götaland County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakellariou G, Conaghan PG, Zhang W, Bijlsma JWJ, Boyesen P, D'Agostino MA, Doherty M, Fodor D, Kloppenburg M, Miese F, Naredo E, Porcheret M, Iagnocco A. EULAR recommendations for the use of imaging in the clinical management of peripheral joint osteoarthritis. Ann Rheum Dis. 2017 Sep;76(9):1484-1494. doi: 10.1136/annrheumdis-2016-210815. Epub 2017 Apr 7. PMID 28389554
- [Background] Ho CM, Thorstensson CA, Nordeman L. Physiotherapist as primary assessor for patients with suspected knee osteoarthritis in primary care-a randomised controlled pragmatic study. BMC Musculoskelet Disord. 2019 Jul 13;20(1):329. doi: 10.1186/s12891-019-2690-1. PMID 31301739
- [Background] Ho-Henriksson CM, Svensson M, Thorstensson CA, Nordeman L. Physiotherapist or physician as primary assessor for patients with suspected knee osteoarthritis in primary care - a cost-effectiveness analysis of a pragmatic trial. BMC Musculoskelet Disord. 2022 Mar 17;23(1):260. doi: 10.1186/s12891-022-05201-3. PMID 35300671
- [Background] Morris L, Moule P, Pearson J, Foster D, Walsh N. Patient acceptability of the physiotherapy first contact practitioner role in primary care: A realist informed qualitative study. Musculoskeletal Care. 2021 Mar;19(1):38-51. doi: 10.1002/msc.1505. Epub 2020 Sep 28. PMID 32989900
- [Background] Goodwin R, Moffatt F, Hendrick P, Timmons S, Chadborn N, Logan P. First point of contact physiotherapy; a qualitative study. Physiotherapy. 2020 Sep;108:29-36. doi: 10.1016/j.physio.2020.02.003. Epub 2020 Feb 19. PMID 32693240
- [Background] Coxon D, Frisher M, Jinks C, Jordan K, Paskins Z, Peat G. The relative importance of perceived doctor's attitude on the decision to consult for symptomatic osteoarthritis: a choice-based conjoint analysis study. BMJ Open. 2015 Oct 26;5(10):e009625. doi: 10.1136/bmjopen-2015-009625. PMID 26503396
- [Background] Miller KA, Osman F, Baier Manwell L. Patient and physician perceptions of knee and hip osteoarthritis care: A qualitative study. Int J Clin Pract. 2020 Dec;74(12):e13627. doi: 10.1111/ijcp.13627. Epub 2020 Aug 11. PMID 32734667
- [Background] Alami S, Boutron I, Desjeux D, Hirschhorn M, Meric G, Rannou F, Poiraudeau S. Patients' and practitioners' views of knee osteoarthritis and its management: a qualitative interview study. PLoS One. 2011 May 5;6(5):e19634. doi: 10.1371/journal.pone.0019634. PMID 21573185
- [Background] Smith TO, Purdy R, Lister S, Salter C, Fleetcroft R, Conaghan PG. Attitudes of people with osteoarthritis towards their conservative management: a systematic review and meta-ethnography. Rheumatol Int. 2014 Mar;34(3):299-313. doi: 10.1007/s00296-013-2905-y. Epub 2013 Dec 5. PMID 24306266
- [Background] Teo PL, Bennell KL, Lawford B, Egerton T, Dziedzic K, Hinman RS. Patient experiences with physiotherapy for knee osteoarthritis in Australia-a qualitative study. BMJ Open. 2021 Mar 8;11(3):e043689. doi: 10.1136/bmjopen-2020-043689. PMID 34006028
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Graneheim UH, Lindgren BM, Lundman B. Methodological challenges in qualitative content analysis: A discussion paper. Nurse Educ Today. 2017 Sep;56:29-34. doi: 10.1016/j.nedt.2017.06.002. Epub 2017 Jun 17. PMID 28651100
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Derived] Ho-Henriksson CM, Thorstensson CA, Nordeman L, Ziden L. "I want to be physically active as long as I live" Expectations and experiences of direct access to physiotherapist in primary healthcare of patients with knee osteoarthritis. Disabil Rehabil. 2026 Feb;48(4):941-950. doi: 10.1080/09638288.2025.2519494. Epub 2025 Jun 17. PMID 40524625
- See also: Swedish national guidelines for musculoskeletal disorders — https://www.socialstyrelsen.se/globalassets/sharepoint-dokument/artikelkatalog/nationella-riktlinjer/2021-1-7137-kunskapsunderlag.pdf